CLINICAL TRIAL: NCT00567528
Title: Comparison of the Efficacy of Topical Ibuprofen to Oral Ibuprofen in Adolescent Athletes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not producing meaningful data.
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Principal Investigator, Eloise Lemon, M.D., Akron Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB #0600210
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2012-01

CONDITIONS: Soft Tissue Injury
Keywords: Soft tissue injuries; Topical ibuprofen; Adolescent athletes
MeSH Terms: conditions — Soft Tissue Injuries | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Active ibuprofen liposomal transdermal gel with placebo ibuprofen capsule
  Interventions: Drug: ibuprofen
- 2 (Other): Placebo ibuprofen liposomal transdermal gel with active ibuprofen capsules
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — Apply by rubbing into skin for 30 to 60 seconds placebo ibuprofen 10% gel, 0.5cc to skin over injured area 3 times a day and taking active capsules of ibuprofen 3 times a day 10-40mg/kg per day, not to exceed 1200mg per day for 2 weeks.
  Arms: 2
Drug: ibuprofen — Apply by rubbing into skin for 30 to 60 seconds active ibuprofen 10% gel, 0.5cc to skin over injured area 3 times a day and taking placebo capsules of ibuprofen 3 times a day 10-40mg/kg per day, not to exceed 1200mg per day for 2 weeks.
  Arms: 1

SUMMARY:
This study was made to compare the efficacy of topical ibuprofen in gel form with oral ibuprofen in the treatment of sub-acute soft tissue injuries while comparing the tolerability of the delivery methods

ELIGIBILITY:
Inclusion Criteria:

* Age 12-19yo
* soft tissue injury or flare up of soft tissue injury within 10 days to 8 weeks

Exclusion Criteria:

* Known hypersensitivity to aspirin or any NSAID,
* allergy to eggs or egg products
* history of asthma, renal disease, GI disease, active or suspected bleeding peptic ulcer (past or present), anemia, hypertension, other systemic disease significantly affecting liver or renal function
* serious injury within six months
* currently on anticoagulants
* pregnant or lactating females
* active arthritis in affected limb
* open wounds, infected skin or fractures
* opioid use within 7 days
* severe psychological disorder
* prior topical medication applied to the painful region/area of study

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2006-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of Topical Ibuprofen to Oral Ibuprofen measured by numeric pain rating, swelling at injury site, and change in sports activity. | 10 days to 8 weeks after initial injury or flare up

SECONDARY OUTCOMES:
Compare the tolerability of the two delivery methods measured by side effects. | 2 weeks after starting topical and oral ibuprofen

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel O Adekunle, M.D., Principal Investigator — Akron Children's Hospital; Joseph Congeni, M.D., Study Director — Akron Children's Hospital; Cynthia Bennett, MSN, CNP, Principal Investigator — Akron Children's Hospital
Locations (1):
- Sports Medicine Department at Akron Children's Hospital, Akron, Ohio, United States

REFERENCES:
- [Background] Whitefield M, O'Kane CJ, Anderson S. Comparative efficacy of a proprietary topical ibuprofen gel and oral ibuprofen in acute soft tissue injuries: a randomized, double-blind study. J Clin Pharm Ther. 2002 Dec;27(6):409-17. doi: 10.1046/j.1365-2710.2002.00439.x. PMID 12472980